CLINICAL TRIAL: NCT02214225
Title: A Phase 3, Randomized, Multicenter, Double-blinded Study to Evaluate the Immunogenicity and Safety of a Quadrivalent Influenza Vaccine (CSL QIV) in Comparison With a US Licensed 2014/2015 Trivalent Influenza Vaccine (CSL TIV-1), and a Trivalent Influenza Vaccine Containing the Alternate B Strain (CSL TIV-2), in Adults Aged 18 Years and Above.
Brief Title: A Study to Evaluate the Immunogenicity and Safety of bioCSL Quadrivalent Influenza Vaccine (QIV) in Adults Aged 18 Years and Above.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-QIV-13-01
Record Dates: First submitted 2014-08-10; First posted 2014-08-12 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Quadrivalent Influenza Vaccine (QIV) (Experimental): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)
- Trivalent Influenza Vaccine (TIV-1) (Active Comparator): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  Interventions: Biological: Trivalent Influenza Vaccine (TIV-1)
- Trivalent Influenza Vaccine (TIV-2) (Active Comparator): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the recommended influenza A (H1N1-, H3N2-like) strains and the alternate B strain for the Northern Hemisphere 2014/2015 influenza season).
  Interventions: Biological: Trivalent Influenza Vaccine (TIV-2)

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (QIV) — One 0.5 mL intramuscular dose into the deltoid muscle
  Arms: Quadrivalent Influenza Vaccine (QIV)
Biological: Trivalent Influenza Vaccine (TIV-1) — One 0.5 mL intramuscular dose into the deltoid muscle.
  Arms: Trivalent Influenza Vaccine (TIV-1)
Biological: Trivalent Influenza Vaccine (TIV-2) — One 0.5 mL intramuscular dose into the deltoid muscle.
  Arms: Trivalent Influenza Vaccine (TIV-2)

SUMMARY:
This is a study to assess the immune (antibody) response and safety of a bioCSL split virion, inactivated quadrivalent influenza vaccine, in comparison with a US licensed 2014/2015 trivalent influenza vaccine (bioCSL TIV-1), and a trivalent influenza vaccine containing the alternate B strain (bioCSL TIV-2), in healthy adult volunteers aged 18 years and above.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blinded study was conducted during the 2014-2015 Northern Hemisphere influenza immunization season to evaluate the non-inferior immune response of bioCSL QIV to that of bioCSL TIV-1 and bioCSL TIV-2 along with safety in healthy male and female adults aged ≥ 18 years. Each vaccinated subject had a maximum 25 day on-study period with a six month safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females aged ≥ 18 years at the time of vaccination.
* Females of child-bearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for the duration of the On-study period. Females of child-bearing potential must return a negative urine pregnancy test result prior to vaccination with the vaccine.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of bioCSL influenza vaccines.
* Vaccination against influenza in the previous 6 months.
* Known history of Guillain-Barré Syndrome or other demyelinating disease.
* Clinical signs of active infection and/or an oral temperature of ≥ 100.4°F (38.0°C).
* A clinically significant medical condition.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3484 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: bioCSL Pty Ltd Clinical Program Director, Study Director — Seqirus
Locations (33):
- United States (33):
  - Site 296, Huntsville, Alabama
  - Site 286, Los Angeles, California
  - Site 315, San Diego, California
  - Site 301, Milford, Connecticut
  - Site 297, Jacksonville, Florida
  - Site 293, Melbourne, Florida
  - Site 292, Savannah, Georgia
  - Site 289, Meridian, Idaho
  - Site 294, Peoria, Illinois
  - Site 295, Mishawaka, Indiana
  - Site 317, Witchita, Kansas
  - Site 291, Rockville, Maryland
  - Site 310, Methuen, Massachusetts
  - Site 287, St Louis, Missouri
  - Site 316, Bellevue, Nebraska
  - Site 298, Las Vegas, Nevada
  - Site 285, Binghamton, New York
  - Site 313, Rochester, New York
  - Site 302, Charlotte, North Carolina
  - Site 306, Raleigh, North Carolina
  - Site 309, Wilmington, North Carolina
  - Site 305, Winston-Salem, North Carolina
  - Site 299, Oklahoma City, Oklahoma
  - Site 307, Mt. Pleasant, South Carolina
  - Site 308, Bristol, Tennessee
  - Site 311, Jefferson City, Tennessee
  - Site 312, Knoxville, Tennessee
  - Site 304, Knoxville, Tennessee
  - Site 283, Austin, Texas
  - Site 282, Forth Worth, Texas
  - Site 288, San Angelo, Texas
  - Site 300, Salt Lake City, Utah
  - Site 303, Charlottesville, Virginia

REFERENCES:
- [Derived] Treanor JT, Albano FR, Sawlwin DC, Graves Jones A, Airey J, Formica N, Matassa V, Leong J. Immunogenicity and safety of a quadrivalent inactivated influenza vaccine compared with two trivalent inactivated influenza vaccines containing alternate B strains in adults: A phase 3, randomized noninferiority study. Vaccine. 2017 Apr 4;35(15):1856-1864. doi: 10.1016/j.vaccine.2017.02.066. Epub 2017 Mar 13. PMID 28302411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 15-AUG-2014, Last Patient Last Visit: 20-APR-2015. Number of activated sites that enrolled subjects: 31 (all based in USA).
Pre-assignment Details: Number of subjects screened: 3673. Number of subjects randomized: 3484.
Groups:
- Quadrivalent Influenza Vaccine (QIV): The study vaccine is a sterile, thiomersal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  Quadrivalent Influenza Vaccine (QIV): One 0.5 mL intramuscular dose into the deltoid muscle
- Trivalent Influenza Vaccine (TIV-1): The study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  Trivalent Influenza Vaccine (TIV-1): One 0.5 mL intramuscular dose into the deltoid muscle.
- Trivalent Influenza Vaccine (TIV-2): The study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the recommended influenza A (H1N1-, H3N2-like) strains and the alternative B strain for the Northern Hemisphere 2014/2015 influenza season).
  Trivalent Influenza Vaccine (TIV-2): One 0.5 mL intramuscular dose into the deltoid muscle.
Period: Overall Study
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2)
Started | 1741 | 871 | 872
Completed | 1686 | 852 | 850
Not Completed | 55 | 19 | 22
Not completed — Lost to Follow-up | 46 | 18 | 18
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Death | 5 | 0 | 1
Not completed — randomized in error, not vaccinated | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was used for analysis of subject characteristics and comprised all subjects who gave informed consent and who were randomized to treatment. Screening failures were not included in the FAS.
Groups:
- Quadrivalent Influenza Vaccine (QIV): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  QIV dose: One 0.5 mL intramuscular dose into the deltoid muscle.
- Trivalent Influenza Vaccine (TIV-1): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  TIV-1 dose: One 0.5 mL intramuscular dose into the deltoid muscle.
- Trivalent Influenza Vaccine (TIV-2): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the recommended influenza A (H1N1-, H3N2-like) strains and the alternative B strain for the Northern Hemisphere 2014/2015 influenza season).
  TIV-2 dose: One 0.5 mL intramuscular dose into the deltoid muscle.
- Total: Total of all reporting groups
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2) | Total
Number analyzed (Participants) | 1741 | 871 | 872 | 3484
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (18.10) | 58.2 (18.10) | 58.3 (17.89) | 58.3 (18.04)
Age, Customized [Number; unit: participants] — Number of participants allocated within each age subset category for each arm.
  participants
    18 to 49 years | 510 | 255 | 255 | 1020
    50 to 64 years | 361 | 179 | 181 | 721
    65 to 74 years | 541 | 271 | 270 | 1082
    => 75 years | 329 | 166 | 166 | 661
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 971 | 511 | 510 | 1992
  Male | 770 | 360 | 362 | 1492
Region of Enrollment [Number; unit: participants]
  United States | 1741 | 871 | 872 | 3484

OUTCOME MEASURES:

1. Primary Outcome: Postvaccination Geometric Mean Titer (GMT) (Statistical Analysis: GMT Ratios) in Subjects Aged ≥18 Years (Per Protocol Population).
Description: Immunogenicity was assessed by measuring HI titers to the four virus strains. Postvaccination GMTs were determined. (GMT dispersion values are based on unadjusted GMT values.) The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was then determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains.
Time Frame: 21 days after vaccination.
Population: The Per Protocol Population was used for the primary and secondary analysis of immunogenicity data and included subjects in the Evaluable Population minus any subjects with deviations that were thought to potentially affect the immunogenicity results, following medical review prior to unblinding.
Measure: Geometric Mean (Full Range); unit: Titer
Groups:
- GMT: bioCSL QIV: Postvaccination GMT.
- GMT: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC): Postvaccination GMT.
  Pooled TIV (A strains), N=1704. TIV-1 (B/YAM), N=854. TIV-2 (B/VIC), N=850.
Arm/Group | GMT: bioCSL QIV | GMT: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC)
Number analyzed (Participants) | 1691 | 1704
Titer
  A/H1N1 | 303.0 [5 to 8127] | 280.2 [5 to 6451]
  A/H3N2 | 488.7 [5 to 10240] | 454.2 [5 to 12902]
  B/Yamagata | 64.3 [5 to 2560] | 55.7 [5 to 2560]
  B/Victoria | 87.9 [5 to 2560] | 82.2 [5 to 5120]
Statistical Analysis 1: Comparison: GMT: bioCSL QIV vs GMT: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); For A/H1N1 strain. The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains; Test type: Non-Inferiority or Equivalence — The non-inferiority criterion for the GMT ratio was that the upper bound of two-sided 95% CI on the ratio of Pooled TIV (for A strains) or TIV-1 (B Yamagata) or TIV-2 (B Victoria)/ bioCSL QIV should not exceed 1.5; GMT ratio (A/H1N1) = 0.92, 95% CI 2-sided [0.87 to 0.98]
Statistical Analysis 2: Comparison: GMT: bioCSL QIV vs GMT: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); For A/H3N2 strain. The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (A/H3N2) = 0.93, 95% CI 2-sided [0.88 to 0.98]
Statistical Analysis 3: Comparison: GMT: bioCSL QIV vs GMT: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); For B/Yamagata strain. The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B/YAM) = 0.87, 95% CI 2-sided [0.81 to 0.93]
Statistical Analysis 4: Comparison: GMT: bioCSL QIV vs GMT: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); For B/Victoria strain. The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B/VIC) = 0.94, 95% CI 2-sided [0.86 to 1.01]

2. Primary Outcome: The Seroconversion Rate (SCR) (Statistical Analysis: Difference in SCR) in Subjects Aged ≥18 Years.
Description: SCR (defined as the percentage of subjects with either a prevaccination HI titer < 1:10 and a postvaccination HI titer ≥ 1:40 or a prevaccination HI titer ≥ 1:10 and a 4-fold increase in postvaccination HI titer) was determined for each virus strain included in the vaccines: bioCSL TIV-1 and bioCSL TIV-2 SCRs were pooled for analysis of the A strains. The SCR difference was defined as the SCR percentage for bioCSL Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus the SCR percentage for bioCSL QIV.
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- SCR: bioCSL QIV: bioCSL QIV, n=1691.
- SCR: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC): Pooled TIV (A strains), n=1704. TIV-1 (B Yamagata), n=854. TIV-2 (B Victoria), n=850.
Arm/Group | SCR: bioCSL QIV | SCR: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC)
Number analyzed (Participants) | 1691 | 1704
percentage of participants
  A/H1N1 | 38.8 | 37.7
  A/H3N2 | 40.9 | 39.3
  B/Yamagata | 31.0 | 27.8
  B/Victoria | 40.3 | 38.7
Statistical Analysis 1: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); Test type: Non-Inferiority or Equivalence — For A/H1N1. The non-inferiority criterion was that the upper bound of the two sided 95% CI on the difference between SCRs (Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus bioCSL QIV) should not exceed 10%; Difference in SCR (A/H1N1) = -1.1, 95% CI 2-sided [-4.4 to 2.2]
Statistical Analysis 2: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); Test type: Non-Inferiority or Equivalence — For A/H3N2. The non-inferiority criterion was that the upper bound of the two sided 95% CI on the difference between SCRs (Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus bioCSL QIV) should not exceed 10%; Difference in SCR (A/H3N2) = -1.7, 95% CI 2-sided [-5.0 to 1.6]
Statistical Analysis 3: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); Test type: Non-Inferiority or Equivalence — For B/Yamagata. The non-inferiority criterion was that the upper bound of the two sided 95% CI on the difference between SCRs (Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus bioCSL QIV) should not exceed 10%; Difference in SCR (B/YAM) = -3.2, 95% CI 2-sided [-7.0 to 0.5]
Statistical Analysis 4: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV (A Strains) or TIV-1 (B/YAM) or TIV-2 (B/VIC); Test type: Non-Inferiority or Equivalence — For B/Victoria. The non-inferiority criterion was that the upper bound of the two sided 95% CI on the difference between SCRs (Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus bioCSL QIV) should not exceed 10%; Difference in SCR (B/VIC) = -1.6, 95% CI 2-sided [-5.6 to 2.4]

3. Secondary Outcome: Postvaccination GMT (Statistical Analyses: GMT Ratios) Assessed Separately Within Each Age Group (18 Through 64 Years and ≥ 65 Years of Age) (Per-Protocol Population).
Description: Immunogenicity was assessed by measuring HI titers to the four virus strains. Postvaccination GMTs were determined. (GMT dispersion values are based on unadjusted GMT values.) The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was then determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains.
  Non-inferiority of bioCSL QIV compared to bioCSL TIV-1, and to bioCSL TIV-2 was assessed separately within each age group (18 to < 65 years and ≥ 65 years of age) through assessment of GMT ratios as described for the primary endpoint.
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Titer
Groups:
- GMT: bioCSL QIV (18 to <65 Years): Postvaccination GMT. bioCSL QIV, n=835.
- GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years): Postvaccination GMT. Pooled TIV (A strains), n=845. TIV-1 (B Yamagata), n=424. TIV-2 (B Victoria), n=421.
- GMT: bioCSL QIV (≥ 65 Years): Postvaccination GMT. bioCSL QIV, n=856.
- GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years): Postvaccination GMT. Pooled TIV (A strains), n=859 TIV-1 (B/YAM), n=430. TIV-2 (B/VIC), n=429.
Arm/Group | GMT: bioCSL QIV (18 to <65 Years) | GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years) | GMT: bioCSL QIV (≥ 65 Years) | GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years)
Number analyzed (Participants) | 835 | 845 | 856 | 859
Titer
  A/H1N1 | 432.7 [10 to 8127] | 402.8 [20 to 6451] | 211.4 [5 to 3225] | 199.8 [5 to 4064]
  A/H3N2 | 569.1 [5 to 10240] | 515.1 [20 to 12902] | 419.5 [5 to 10240] | 400.0 [5 to 5120]
  B/Yamagata | 92.3 [5 to 2560] | 79.3 [5 to 2560] | 43.3 [5 to 1613] | 39.1 [5 to 1280]
  B/Victoria | 110.7 [10 to 2560] | 95.2 [5 to 5120] | 66.1 [5 to 2560] | 68.4 [5 to 2560]
Statistical Analysis 1: Comparison: GMT: bioCSL QIV (18 to <65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (A/H1N1) = 0.93, 95% CI 2-sided [0.85 to 1.02]
Statistical Analysis 2: Comparison: GMT: bioCSL QIV (18 to <65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (A/H3N2) = 0.91, 95% CI 2-sided [0.83 to 0.99]
Statistical Analysis 3: Comparison: GMT: bioCSL QIV (18 to <65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); For B/YAM strain. The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B/YAM) = 0.86, 95% CI 2-sided [0.76 to 0.97]
Statistical Analysis 4: Comparison: GMT: bioCSL QIV (18 to <65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); For B/VIC strain. The GMT ratio (defined as the geometric mean of postvaccination (day 21) HI titer for TIV divided by the geometric mean of the postvaccination HI titer for QIV) for each virus strain included in the vaccines was determined: bioCSL TIV-1 and bioCSL TIV-2 GMTs were pooled for analysis of the A strains; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B/VIC) = 0.86, 95% CI 2-sided [0.76 to 0.98]
Statistical Analysis 5: Comparison: GMT: bioCSL QIV (≥ 65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (A/H1N1) = 0.95, 95% CI 2-sided [0.88 to 1.02]
Statistical Analysis 6: Comparison: GMT: bioCSL QIV (≥ 65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (A/H3N2) = 0.95, 95% CI 2-sided [0.89 to 1.02]
Statistical Analysis 7: Comparison: GMT: bioCSL QIV (≥ 65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 3, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B/YAM) = 0.90, 95% CI 2-sided [0.84 to 0.97]
Statistical Analysis 8: Comparison: GMT: bioCSL QIV (≥ 65 Years) vs GMT: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 3, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B/VIC) = 1.03, 95% CI 2-sided [0.94 to 1.14]

4. Secondary Outcome: The Seroconversion Rate (SCR) (Statistical Analyses: Difference in SCR) for Each Virus Strain, Assessed Separately Within Each Age Group (18 to < 65 Years and ≥ 65 Years of Age) (Per Protocol Population).
Description: Non-inferiority of bioCSL QIV compared to bioCSL TIV-1, and to bioCSL TIV-2 was assessed separately within each age group (18 to < 65 years and ≥ 65 years of age) through assessment of SCR differences as described for the primary endpoint.
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Groups:
- SCR: bioCSL QIV (18 to < 65 Years): bioCSL TIV-1 and bioCSL TIV-2 are pooled for analysis of the A strains. For B/Yamagata TIV=TIV-1, for B/Victoria TIV=TIV-2.
  bioCSL QIV, n=835. Pooled TIV (A strains), n=845. TIV-1 (B Yamagata), n=424. TIV-2 (B Victoria), n=421.
- SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); SCR: bioCSL QIV (≥ 65 Years); SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years): bioCSL TIV-1 and bioCSL TIV-2 are pooled for analysis of the A strains. For B/Yamagata TIV=TIV-1, for B/Victoria TIV=TIV-2.
  bioCSL QIV, n=856. Pooled TIV (A strains), n=859. TIV-1 (B Yamagata), n=430. TIV-2 (B Victoria), n=429.
Arm/Group | SCR: bioCSL QIV (18 to < 65 Years) | SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years) | SCR: bioCSL QIV (≥ 65 Years) | SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years)
Number analyzed (Participants) | 835 | 845 | 856 | 859
percentage of participants analyzed
  A/H1N1 | 51.3 | 49.1 | 26.6 | 26.4
  A/H3N2 | 56.3 | 51.7 | 25.9 | 27.0
  B/Yamagata | 45.7 | 41.3 | 16.6 | 14.4
  B/Victoria | 57.6 | 53.0 | 23.5 | 24.7
Statistical Analysis 1: Comparison: SCR: bioCSL QIV (18 to < 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); The SCR difference was defined as the SCR percentage for bioCSL Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus the SCR percentage for bioCSL QIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in SCR (A/H1N1) = -2.1, 95% CI 2-sided [-6.9 to 2.6]
Statistical Analysis 2: Comparison: SCR: bioCSL QIV (18 to < 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Difference in SCR (A/H3N2) = -4.6, 95% CI 2-sided [-9.3 to 0.2]
Statistical Analysis 3: Comparison: SCR: bioCSL QIV (18 to < 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — For B/YAM. The non-inferiority criterion was that the upper bound of the two sided 95% CI on the difference between SCRs (Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus bioCSL QIV) should not exceed 10%; Difference in SCR (B/YAM) = -4.5, 95% CI 2-sided [-10.3 to 1.3]
Statistical Analysis 4: Comparison: SCR: bioCSL QIV (18 to < 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (18 to <65years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — For B/VIC. The non-inferiority criterion was that the upper bound of the two sided 95% CI on the difference between SCRs (Pooled TIV or TIV-1 (B Yamagata) or TIV-2 (B Victoria) minus bioCSL QIV) should not exceed 10%; Difference in SCR (B/VIC) = -4.6, 95% CI 2-sided [-10.5 to 1.2]
Statistical Analysis 5: Comparison: SCR: bioCSL QIV (≥ 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in SCR (A/H1N1) = -0.2, 95% CI 2-sided [-4.4 to 4.0]
Statistical Analysis 6: Comparison: SCR: bioCSL QIV (≥ 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Difference in SCR (A/H3N2) = 1.1, 95% CI 2-sided [-3.1 to 5.2]
Statistical Analysis 7: Comparison: SCR: bioCSL QIV (≥ 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 3]; Difference in SCR (B/YAM) = -2.2, 95% CI 2-sided [-6.3 to 2.0]
Statistical Analysis 8: Comparison: SCR: bioCSL QIV (≥ 65 Years) vs SCR: Pooled TIV (A Strains) or TIV-1 or TIV-2 (≥ 65 Years); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 4]; Difference in SCR (B/VIC) = 1.2, 95% CI 2-sided [-3.7 to 6.2]

5. Secondary Outcome: Immunologic Superiority of the Alternate B Strain in bioCSL QIV, as Determined by the GMT (Statistical Analysis: GMT Ratio) for This Strain, Overall and by Age Cohort (Per Protocol Population).
Description: Immunologic superiority of the alternate B strain (ie, the influenza B strain included in the QIV but not in the TIV formulation) in bioCSL QIV was assessed separately within each age group (18 to < 65 years and ≥ 65 years of age), and overall. The GMT ratio was calculated as bioCSL QIV GMT/bioCSL TIV GMT for the superiority analyses, which is the reverse of how it was calculated for the non-inferiority analyses.
  (GMT dispersion values are based on unadjusted GMT values.)
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Titer
Groups:
- Postvaccination GMT: bioCSL QIV: bioCSL QIV, Adults 18 years and older, N=1691. 18 to < 65 years, n=835. => 65 years, n=856.
- Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC): B/Yamagata serology for TIV-2 (B Victoria), Adults 18 years and older, n=850 B/Victoria serology for TIV-1 (B Yamagata), Adults 18 years and older, n=854 B/Yamagata serology for TIV-2 (B Victoria), Adults 18 through 64 years inclusive, n=421 B/Victoria serology for TIV-1 (B Yamagata), Adults 18 through 64 years inclusive, n=424 B/Yamagata serology for TIV-2 (B Victoria), Adults 65 years and older, n=429 B/Victoria serology for TIV-1 (B Yamagata), Adults 65 years and older, n=430.
Arm/Group | Postvaccination GMT: bioCSL QIV | Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC)
Number analyzed (Participants) | 1691 | 854
Titer
  B/Yamagata (overall, ≥18 years) | 62.9 [5 to 2560] | 42.7 [5 to 2560]
  B/Victoria (overall, ≥18 years) | 86.9 [5 to 2560] | 55.4 [5 to 5120]
  B/Yamagata (18 to <65 years) | 89.9 [5 to 2560] | 53.8 [5 to 2560]
  B/Victoria (18 to <65 years) | 113.5 [10 to 2560] | 64.3 [5 to 5120]
  B/Yamagata (≥65 years) | 43.8 [5 to 1613] | 33.6 [5 to 1280]
  B/Victoria (≥65 years) | 64.1 [5 to 2560] | 46.3 [5 to 2560]
Statistical Analysis 1: Comparison: Postvaccination GMT: bioCSL QIV vs Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC); Immunologic superiority of the alternate B strain (ie, the influenza B strain included in the QIV but not in the TIV formulation) in bioCSL QIV was assessed separately within each age group (18 to < 65 years and ≥ 65 years of age), and overall. The GMT ratio was calculated as bioCSL QIV GMT/bioCSL TIV GMT for the superiority analyses, which is the reverse of how it was calculated for the non-inferiority analyses; Test type: Superiority or Other; GMT ratio (B/YAM) overall = 1.47, 95% CI 2-sided [1.38 to 1.57] — Immunologic superiority of the alternate B strain (eg, the influenza B strain included in the bioCSL QIV but not in the bioCSL TIV formulation) in bioCSL QIV was demonstrated if the lower bound of the two-sided 95% CI on GMT ratio was greater than 1
Statistical Analysis 2: Comparison: Postvaccination GMT: bioCSL QIV vs Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; GMT ratio (B/VIC) overall = 1.57, 95% CI 2-sided [1.45 to 1.70] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Postvaccination GMT: bioCSL QIV vs Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; GMT ratio (B/YAM) 18 through 64 years = 1.67, 95% CI 2-sided [1.50 to 1.87] — Immunologic superiority of the alternate B strain (eg, the influenza B strain included in the bioCSL QIV but not in the bioCSL TIV formulation) in bioCSL QIV was demonstrated if the lower bound of the two-sided 95% CI on GMT was greater than 1
Statistical Analysis 4: Comparison: Postvaccination GMT: bioCSL QIV vs Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; GMT ratio (B/VIC) 18 through 64 years = 1.76, 95% CI 2-sided [1.55 to 2.01] — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 5: Comparison: Postvaccination GMT: bioCSL QIV vs Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; GMT ratio (B/YAM) ≥ 65 years = 1.30, 95% CI 2-sided [1.21 to 1.40] — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 6: Comparison: Postvaccination GMT: bioCSL QIV vs Postvaccination GMT: TIV-1 (B/YAM) or TIV-2 (B/VIC); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; GMT ratio (B/VIC) ≥ 65 years = 1.38, 95% CI 2-sided [1.27 to 1.51] — [estimate comment as in outcome 5, analysis 3]

6. Secondary Outcome: Immunologic Superiority of the Alternate B Strain in bioCSL QIV, as Determined by Seroconversion Rate (SCR) (Statistical Analysis: Difference in SCR) for This Strain, Overall and by Age Cohort (Per Protocol Population)
Description: Immunologic superiority of the alternate B strain (ie, the influenza B strain included in the QIV but not in the TIV formulation) in bioCSL QIV was assessed separately within each age group (18 to < 65 years and ≥ 65 years of age), and overall. The SCR difference was calculated as bioCSL QIV SCR minus bioCSL TIV SCR, which is the reverse of how it was calculated for the non-inferiority analyses. For the SCR comparison superiority was demonstrated if the lower limit of the two-sided 95% CI of the difference of the seroconversion rates was greater than 0 for each B strain in QIV compared with the corresponding B strain not contained in each TIV.
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Number; unit: percentage of participants analyzed
Groups:
- SCR: bioCSL QIV: For B/Yamagata TIV=TIV-1, for B/Victoria TIV=TIV-2.
  bioCSL QIV, Adults 18 years and older, n=1691. bioCSL QIV, Adults 18 years to <65 years, n=835. bioCSL QIV, Adults 65 years and older, n=856.
- SCR: Pooled TIV-1 or TIV-2: For B/Yamagata TIV=TIV-1, for B/Victoria TIV=TIV-2.
  B/Yamagata serology for TIV-2 (B Victoria), Adults 18 years and older, n=850. B/Victoria serology for TIV-1 (B Yamagata), Adults 18 years and older, n=854. B/Yamagata serology for TIV-2 (B Victoria), Adults 18 to <65 years, n=421. B/Victoria serology for TIV-1 (B Yamagata), Adults 18 years to <65 years, n=424.
  B/Yamagata serology for TIV-2 (B Victoria), Adults 65 years and older, n=429. B/Victoria serology for TIV-1 (B Yamagata), Adults 65 years and older, n=430.
Arm/Group | SCR: bioCSL QIV | SCR: Pooled TIV-1 or TIV-2
Number analyzed (Participants) | 1691 | 854
percentage of participants analyzed
  B/Yamagata (overall, ≥18 years) | 31.0 | 15.6
  B/Victoria (overall, ≥18 years) | 40.3 | 20.3
  B/Yamagata (18 to <65 years) | 45.7 | 22.8
  B/Victoria (18 to <65 years) | 57.6 | 29.0
  B/Yamagata (≥65 years) | 16.6 | 8.6
  B/Victoria (≥65 years) | 23.5 | 11.6
Statistical Analysis 1: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV-1 or TIV-2; Immunologic superiority of the alternate B strain (ie, the influenza B strain included in the QIV but not in the TIV formulation) in bioCSL QIV was assessed separately within each age group (18 to < 65 years and ≥ 65 years of age), and overall. Seroconversion rate difference = bioCSL QIV SCR percentage - bioCSL TIV-1 or TIV-2 SCR percentage; Test type: Superiority or Other; Difference in SCR (B/YAM) overall = 15.3, 95% CI 2-sided [12.1 to 18.6] — Immunologic superiority of the alternate B strain (eg, the influenza B strain included in bioCSL QIV but not in the TIV formulation) in bioCSL QIV was demonstrated if the lower bound of the two-sided 95% CI for the difference in SCRs was > 0
Statistical Analysis 2: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV-1 or TIV-2; Seroconversion rate difference = bioCSL QIV SCR percentage - bioCSL TIV-1 or TIV-2 SCR percentage; Test type: Superiority or Other; Difference in SCR (B/VIC) overall = 20.1, 95% CI 2-sided [16.5 to 23.6] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV-1 or TIV-2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Difference in SCR (B/YAM) 18 through 64y = 22.9, 95% CI 2-sided [17.7 to 28.2] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV-1 or TIV-2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Difference in SCR (B/VIC) 18 through 64y = 28.6, 95% CI 2-sided [23.1 to 34.1] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV-1 or TIV-2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Difference in SCR (B/YAM) ≥ 65 years = 8.0, 95% CI 2-sided [4.3 to 11.6] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: SCR: bioCSL QIV vs SCR: Pooled TIV-1 or TIV-2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Difference in SCR (B/VIC) ≥ 65 years = 11.9, 95% CI 2-sided [7.7 to 16.0] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Geometric Mean of HI Titers (GMTs) Prevaccination and Postvaccination.
Description: The immunogenicity of bioCSL QIV, bioCSL TIV-1 and bioCSL TIV-2 was assessed in terms of geometric mean HI titers (GMT) prevaccination (Day 1) and postvaccination (Day 21), in age cohorts (per protocol population).
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | bioCSL QIV (18 to <65 Years) | bioCSL TIV-1 (B/YAM) (18 to <65 Years) | bioCSL TIV-2 (B/VIC) (18 to <65 Years) | bioCSL QIV (≥ 65 Years) | bioCSL TIV-1 (B/YAM) (≥ 65 Years) | bioCSL TIV-2 (B/VIC) (≥ 65 Years)
Number analyzed (Participants) | 835 | 424 | 421 | 856 | 430 | 429
Titer
  A/H1N1 (pre-vaccination) | 78.1 [70.51 to 86.41] | 82.3 [71.57 to 94.74] | 82.8 [71.98 to 95.17] | 75.7 [69.93 to 81.84] | 72.0 [64.58 to 80.25] | 69.2 [61.91 to 77.27]
  A/H3N2 (pre-vaccination) | 97.4 [87.93 to 107.96] | 96.1 [83.51 to 110.64] | 105.7 [92.63 to 120.53] | 153.0 [141.90 to 165.05] | 139.0 [123.74 to 156.16] | 142.7 [126.73 to 160.75]
  B/Yamagata (pre-vaccination) | 23.7 [21.89 to 25.61] | 24.7 [22.09 to 27.60] | 23.7 [21.32 to 26.42] | 20.3 [19.01 to 21.70] | 18.6 [17.02 to 20.35] | 19.6 [17.77 to 21.72]
  B/Victoria (pre-vaccination) | 20.4 [18.95 to 21.85] | 20.4 [18.49 to 22.56] | 21.7 [19.54 to 24.04] | 24.4 [22.84 to 26.17] | 23.4 [21.31 to 25.73] | 25.1 [22.73 to 27.63]
  A/H1N1 (post-vaccination) | 429.9 [400.38 to 461.61] | 432.8 [392.96 to 476.66] | 433.9 [391.46 to 481.01] | 175.9 [163.61 to 189.11] | 169.3 [152.67 to 187.68] | 158.7 [143.15 to 175.95]
  A/H3N2 (post-vaccination) | 533.3 [496.04 to 573.37] | 499.4 [449.73 to 554.62] | 532.5 [482.62 to 587.64] | 356.4 [333.25 to 381.14] | 336.6 [305.26 to 371.11] | 330.3 [297.27 to 367.07]
  B/Yamagata (post-vaccination) | 97.4 [90.04 to 105.35] | 84.6 [75.64 to 94.65] | 53.5 [47.85 to 59.88] | 38.1 [35.50 to 40.86] | 33.2 [30.18 to 36.51] | 28.6 [25.75 to 31.69]
  B/Victoria (post-vaccination) | 111.9 [103.57 to 120.82] | 55.5 [49.85 to 61.77] | 103.0 [92.38 to 114.78] | 54.0 [49.97 to 58.40] | 38.7 [34.96 to 42.92] | 57.4 [51.34 to 64.29]

8. Secondary Outcome: Geometric Mean Fold Titer Change From Prevaccination to Postvaccination.
Description: The immunogenicity of bioCSL QIV, bioCSL TIV-1 and bioCSL TIV-2 assessed in terms of Geometric Mean Fold Increase (GMFI, defined as the geometric mean of the fold increases of postvaccination antibody titer over the prevaccination antibody titer) by Age Cohort (Per Protocol Population).
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change Titer (GMFI)
Arm/Group | bioCSL QIV (18 to <65 Years) | bioCSL TIV-1 (B/YAM) (18 to <65 Years) | bioCSL TIV-2 (B/VIC) (18 to <65 Years) | bioCSL QIV (≥ 65 Years) | bioCSL TIV-1 (B/YAM) (≥ 65 Years) | bioCSL TIV-1 (B/VIC) (≥ 65 Years)
Number analyzed (Participants) | 835 | 424 | 421 | 856 | 430 | 429
Fold Change Titer (GMFI)
  A/H1N1 | 5.5 [4.96 to 6.11] | 5.3 [4.53 to 6.10] | 5.2 [4.49 to 6.12] | 2.3 [2.18 to 2.48] | 2.4 [2.14 to 2.58] | 2.3 [2.09 to 2.52]
  A/H3N2 | 5.5 [4.98 to 6.02] | 5.2 [4.56 to 5.91] | 5.0 [4.43 to 5.74] | 2.3 [2.19 to 2.47] | 2.4 [2.21 to 2.65] | 2.3 [2.10 to 2.55]
  B/Yamagata | 4.1 [3.78 to 4.47] | 3.4 [3.05 to 3.85] | 2.3 [2.08 to 2.45] | 1.9 [1.79 to 1.97] | 1.8 [1.67 to 1.91] | 1.5 [1.38 to 1.54]
  B/Victoria | 5.5 [5.04 to 5.99] | 2.7 [2.46 to 3.00] | 4.8 [4.21 to 5.36] | 2.2 [2.08 to 2.34] | 1.7 [1.54 to 1.77] | 2.3 [2.10 to 2.50]

9. Secondary Outcome: Seroprotection Rates Prevaccination and Postvaccination.
Description: The immunogenicity of bioCSL QIV, bioCSL TIV-1 and bioCSL TIV-2 was assessed in terms of percentage of subjects with a HI titer ≥40 (seroprotection rates) prevaccination (Day 1) and postvaccination (Day 21), in age cohorts (per protocol population).
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | bioCSL QIV (18 to <65 Years) | bioCSL TIV-1 (B/YAM) (18 to <65 Years) | bioCSL TIV-2 (B/VIC) (18 to <65 Years) | bioCSL QIV (≥ 65 Years) | bioCSL TIV-1 (B/YAM) (≥ 65 Years) | bioCSL TIV-1 (B/VIC) (≥ 65 Years)
Number analyzed (Participants) | 835 | 424 | 421 | 856 | 430 | 429
percentage of participants
  A/H1N1 (pre-vaccination) | 73.2 [70.0 to 76.2] | 76.9 [72.6 to 80.8] | 75.5 [71.1 to 79.6] | 78.5 [75.6 to 81.2] | 80.0 [75.9 to 83.7] | 77.4 [73.1 to 81.3]
  A/H3N2 (pre-vaccination) | 78.3 [75.4 to 81.1] | 77.1 [72.8 to 81.0] | 81.5 [77.4 to 85.1] | 92.9 [90.9 to 94.5] | 90.9 [87.8 to 93.5] | 88.8 [85.4 to 91.6]
  B/Yamagata (pre-vaccination | 39.9 [36.5 to 43.3] | 39.9 [35.2 to 44.7] | 40.9 [36.1 to 45.7] | 33.2 [30.0 to 36.4] | 29.1 [24.8 to 33.6] | 31.2 [26.9 to 35.9]
  B/Victoria (pre-vaccination) | 33.5 [30.3 to 36.8] | 32.8 [28.3 to 37.5] | 35.9 [31.3 to 40.7] | 38.7 [35.4 to 42.0] | 36.3 [31.7 to 41.0] | 40.1 [35.4 to 44.9]
  A/H1N1 (post-vaccination) | 99.0 [98.1 to 99.6] | 100.0 [99.1 to 100.0] | 99.0 [97.6 to 99.7] | 94.6 [92.9 to 96.0] | 95.8 [93.5 to 97.5] | 95.3 [92.9 to 97.1]
  A/H3N2 (post-vaccination) | 99.0 [98.1 to 99.6] | 98.8 [97.3 to 99.6] | 98.8 [97.3 to 99.6] | 99.8 [99.2 to 100.0] | 99.1 [97.6 to 99.7] | 98.1 [96.4 to 99.2]
  B/Yamagata (post-vaccination) | 84.3 [81.7 to 86.7] | 81.4 [77.3 to 85.0] | 68.4 [63.7 to 72.8] | 57.5 [54.1 to 60.8] | 54.2 [49.3 to 59.0] | 46.2 [41.4 to 51.0]
  B/Victoria (post-vaccination) | 86.7 [84.2 to 88.9] | 68.2 [63.5 to 72.6] | 86.2 [82.6 to 89.4] | 68.3 [65.1 to 71.4] | 54.4 [49.6 to 59.2] | 68.3 [63.7 to 72.7]

10. Secondary Outcome: Seroconversion Rates
Description: The immunogenicity of bioCSL QIV, bioCSL TIV-1 and bio CSL TIV-2 was assessed in terms of the seroconversion rate, ie, percentage of subjects with either a prevaccination HI titer < 1:10 and a postvaccination HI titer ≥ 1:40, or a prevaccination titer ≥ 1:10 and a ≥ 4-fold increase in post-vaccination titer. Data presented in age cohorts (per protocol population).
Time Frame: 21 days after vaccination.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | bioCSL QIV (18 to <65 Years) | bioCSL TIV-1 (B/YAM) (18 to <65 Years) | bioCSL TIV-2 (B/VIC) (18 to <65 Years) | bioCSL QIV (≥ 65 Years) | bioCSL TIV-1 (B/YAM) (≥ 65 Years) | bioCSL TIV-1 (B/VIC) (≥ 65 Years)
Number analyzed (Participants) | 835 | 424 | 421 | 856 | 430 | 429
percentage of participants
  A/H1N1 | 51.3 [47.8 to 54.7] | 50.5 [45.6 to 55.3] | 47.7 [42.9 to 52.6] | 26.6 [23.7 to 29.7] | 27.4 [23.3 to 31.9] | 25.4 [21.4 to 29.8]
  A/H3N2 | 56.3 [52.8 to 59.7] | 52.8 [48.0 to 57.7] | 50.6 [45.7 to 55.5] | 25.9 [23.0 to 29.0] | 28.6 [24.4 to 33.1] | 25.4 [21.4 to 29.8]
  B/Yamagata | 45.7 [42.3 to 49.2] | 41.3 [36.5 to 46.1] | 22.8 [18.9 to 27.1] | 16.6 [14.2 to 19.3] | 14.4 [11.2 to 18.1] | 8.6 [6.1 to 11.7]
  B/Victoria | 57.6 [54.2 to 61.0] | 29.0 [24.7 to 33.6] | 53.0 [48.1 to 57.8] | 23.5 [20.7 to 26.5] | 11.6 [8.8 to 15.0] | 24.7 [20.7 to 29.1]

11. Secondary Outcome: The Frequency and Severity of Solicited Local and Systemic Adverse Events (AEs).
Description: The overall number of subjects experiencing at least one event of a local and systemic solicited AE, and the overall number of subjects with at least one severe (grade 3) local and systemic solicited AE.
Time Frame: For 7 days following vaccination.
Population: The Safety Population was used for the analysis of safety and comprised all subjects in the Full Analysis Set (FAS) who received the study vaccine and provided follow-up safety data. A statement that they were no AEs constituted follow-up safety data. A total of 31 subjects were assessed as having no follow-up safety data post-vaccination.
Measure: Number; unit: participants
Groups:
- Trivalent Influenza Vaccine (TIV-2): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the recommended influenza A (H1N1-, H3N2-like) strains and the alternative B strain for the Northern Hemisphere 2014/2015 influenza season).
  Trivalent Influenza Vaccine (TIV-2): One 0.5 mL intramuscular dose into the deltoid muscle.
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2)
Number analyzed (Participants) | 1721 | 864 | 864
participants
  Frequency of solicited AEs | 803 | 391 | 397
  Severe (grade 3) solicited AEs | 42 | 15 | 24

12. Secondary Outcome: The Frequency of Cellulitis-like Reaction and Cellulitis.
Description: The number of subjects experiencing at least one episode of each event.
Time Frame: For 28 days following vaccination.
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2)
Number analyzed (Participants) | 1721 | 864 | 864
participants | 0 | 0 | 0

13. Secondary Outcome: The Frequency and Severity of Unsolicited AEs.
Description: The overall number of subjects experiencing at least one event of an unsolicited AE, and the overall number of subjects with at least one severe (grade 3) unsolicited AE.
Time Frame: For 28 days following vaccination.
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2)
Number analyzed (Participants) | 1721 | 864 | 864
participants
  At least one unsolicited AE | 351 | 191 | 176
  Severe (grade 3) unsolicited AE | 73 | 29 | 33

14. Secondary Outcome: The Frequency of Serious Adverse Events (SAEs) for 6 Months Following Vaccination.
Description: The number of participants reporting Serious Adverse Events for 6 months following vaccination.
Time Frame: For 6 months following vaccination.
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2)
Number analyzed (Participants) | 1721 | 864 | 864
participants | 39 | 14 | 13

ADVERSE EVENTS:
Time Frame: Local and systemic solicited AEs collected from Day 1 to Day 7. Unsolicited AEs collected for 28 days after vaccination. SAEs collected for 6 months after vaccination.
Description: The Safety Population was used for the analysis of safety and comprised all subjects in the Full Analysis Set (FAS) who received the study vaccine and provided follow-up safety data. A statement that they were no AEs constituted follow-up safety data. A total of 31 subjects were assessed as having no follow-up safety data post-vaccination.
Arm/Group | Quadrivalent Influenza Vaccine (QIV) | Trivalent Influenza Vaccine (TIV-1) | Trivalent Influenza Vaccine (TIV-2)
Serious Adverse Events (participants affected / at risk) | 39/1721 | 14/864 | 13/864
Other Adverse Events (participants affected / at risk) | 872/1721 | 445/864 | 397/864
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Influenza Vaccine (QIV) (N=1721) | Trivalent Influenza Vaccine (TIV-1) (N=864) | Trivalent Influenza Vaccine (TIV-2) (N=864)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spasmodic dysphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Esophageal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postprocedural hematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abominable pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Influenza Vaccine (QIV) (N=1721) | Trivalent Influenza Vaccine (TIV-1) (N=864) | Trivalent Influenza Vaccine (TIV-2) (N=864)
Pain (General disorders) | 622 (629) | 286 (292) | 309 (316)
Headache (Nervous system disorders) | 258 (300) | 96 (113) | 116 (133)
Malaise (Nervous system disorders) | 114 (125) | 61 (67) | 62 (72)
Myalgia (Musculoskeletal and connective tissue disorders) | 328 (352) | 161 (171) | 157 (173)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
bioCSL agreements and restrictions on publishing may vary with individual investigators; however, bioCSL will not prohibit any investigator from publishing. bioCSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.

(Note: bioCSL was previously known as CSL Biotherapies; bioCSL QIV & TIV were called CSL QIV & TIV in the original protocol)